CLINICAL TRIAL: NCT04951531
Title: Allogeneic Bone-patellar Tendon-bone Transplantation to Reconstruct the Knee Joint Anterior Cruciate Ligament
Brief Title: Allogeneic Bone-patellar Tendon-bone Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200506A
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BPTB double-bundle allograft group (Experimental): The patient underwent arthroscopic double-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) allograft．
  Interventions: Procedure: BPTB double-bundle allograft
- BPTB single-bundle allograft group (Active Comparator): The patient underwent arthroscopic single-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) allograft．
  Interventions: Procedure: BPTB single-bundle allograft group
- BPTB single-bundle autograft group (Active Comparator): The patient underwent arthroscopic single-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) autograft．
  Interventions: Procedure: BPTB single-bundle autograft group

INTERVENTIONS:
Procedure: BPTB double-bundle allograft — The patient underwent surgery of arthroscopic double-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) allograft．
  Arms: BPTB double-bundle allograft group
Procedure: BPTB single-bundle allograft group — The patient underwent surgery of arthroscopic single-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) allograft．
  Arms: BPTB single-bundle allograft group
Procedure: BPTB single-bundle autograft group — The patient underwent surgery of arthroscopic single-bundle anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone (BPTB) autograft．
  Arms: BPTB single-bundle autograft group

SUMMARY:
Objective To investigate the mid-term clinical effect of bone-patellar tendon-bone (BPTB) graft double-bundle reconstruction of the anterior cruciate ligament (ACL) of the knee joint under arthroscope.

DETAILED DESCRIPTION:
The purpose of the present study was to report a unique technique of Double-bundle anterior cruciate ligament reconstruction (DB-ACLR) with a bone-patellar tendon- bone (BPTB) allograftand compare the clinical outcome of the new technique with that of the nonanatomic conventional transtibial Single-bundle anterior cruciate ligament reconstruction (SB-ACLR) with a BPTB allograft. The hypothesis was that the DB-ACLR with a BPTB allograft is technically feasible and may be superior in restoring anterior and rotational stability of the knee joint. Meanwhile, the back-pushing KT- 2000 arthrometer was used to confirm whether there were advantages of DB-ACLR in total anteroposterior stability.

ELIGIBILITY:
Inclusion Criteria:

From July 2005 to June 2008, 3757 ACLRs were performed in our department. A total of 111 patients chose to use allografts, and the other patients chose autologous semitendinosus and gracilis tendons (STGs). The patients selected DB or SB reconstruction based on their understanding about the information from the surgeons. Following the criteria of a prospective randomized study, 56 patients undergoing ACLRs with BPTB allografts were included in our study and were divided into a DB group and a SB group, each with 28 patients. 25 DB and 27 SB patients completed the final follow-up. Only patients between 16 and 50 years old who were undergoing primary operation were included, and younger patients had to have radiographic confirmation of a closed epiphysis.

Exclusion Criteria:

The exclusion criteria included age more than 50 years, narrow middle intercondylar width (<12 mm measured during operation with the knee flexed to 90°), revision reconstruction, multiligament injury, bilateral ACLRs, total meniscectomy or more than one-third partial meniscectomy, and severe cartilage injury.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
side-to-side difference | Before and 2 to 5 years after the operation
  The side-to-side difference was measured at final follow-up by KT-2000 arthrometer (MEDmetric, San Diego, California) at 15 lb, 20 lb, and 30 lb in 30° and 90° of flexion.
total anteroposterior (AP) laxity | Before and 2 to 5 years after the operation
  the total AP laxity (by back-pushing KT-2000 arthrometer measurement) of the knee joint were measured. The technique of the back-pushing KT-2000 arthrometer is as follows: at 30° or 90° of flexion, the patient relaxed himself or herself; next, the examiner pushed back the handle of the KT-2000 arthrometer with 20-lb force and set the zero point of the arthrometer while the tibia was kept in a back position. Then, the examiner applied an anterior force of 15 lb, 20 lb, and 30 lb, respectively, and recorded the results as the total AP laxity of the knee joint.
pivot shift | Before and 2 to 5 years after the operation
  The pivot shift test of the knee joint is a test with an accuracy of 99% in the detection of knee anterior cruciate ligament injury.
range of motion (ROM) | Before and 2 to 5 years after the operation
  Knee joint range of motion. Normal flexion 0 to 130°, extension 0°, flexion internal rotation 0 to 30°, flexion external rotation 0 to 40°.
isokinetic muscle strength evaluation | Before and 2 to 5 years after the operation
  muscle strength was evaluated by Biodex dynamometer (Biodex, Shirley, New York) according to the manufacturer's guidelines. Strength testing was performed for knee flexion and knee extension at 60 and 120 deg/s. The mean peak torque of 5 maximal repetitions for each velocity was assessed to analyze the quadriceps and hamstring isokinetic strength, and the results of the operated leg were expressed as a percentage of that of the nonoperated side.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | Before and 2 to 5 years after the operation
  At present, it is recognized internationally that IKDC has relatively high reliability, effectiveness and sensitivity for the assessment of ligament injuries, especially anterior cruciate ligament injuries.
Tegner score | Before and 2 to 5 years after the operation
  This score is widely used by exercise assessors for patients with knee joint disease. This scoring method divides the patient's exercise level into 0-10 points, 0 as disability, and 10 as being able to participate in national competitive sports.
Lysholm score | Before and 2 to 5 years after the operation
  This score is often used together with the Tegner score. The scores of this scoring system are generally high and focus more on the assessment of daily activities rather than sports.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Prof., Study Chair — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No